CLINICAL TRIAL: NCT04870515
Title: TRIPLE-A PILOT: Actively Intercepting ADT-Induced Metabolic Aberrations in Newly Diagnosed Prostate Cancer
Brief Title: Diet and Physical Activity Intervention for the Prevention of ADT-Induced Metabolic Changes in Patients With Prostate Cancer, TRIPLE-A PILOT Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Marian Neuhouser, Professor, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RG1121348; NCI-2021-02762 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P50CA097186 (NIH); 10669 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2021-04-19; First posted 2021-05-03 (Actual); Results first posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Localized Prostate Carcinoma; Prostate Adenocarcinoma
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care; Diet Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (diet, physical activity) (Experimental): Patients attend 10 in-person or virtual sessions with a registered dietitian over 6 months to receive instruction on healthy dietary pattern. Patients also attend 2 one-on-one sessions with an exercise physiologist to receive instruction on aerobic physical activity and strength/resistance training. Patients may also complete up to 21 additional supervised exercise sessions.
  Interventions: Other: Dietary Intervention; Other: Exercise Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group II (standard lifestyle recommendations) (Active Comparator): Patients attend a single session with a dietitian to review healthy lifestyle recommendations, including US dietary guidelines and 30 minutes of physical activity 5 days/week.
  Interventions: Other: Best Practice; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive standard lifestyle recommendations
  Other Names: standard of care; standard therapy
  Arms: Group II (standard lifestyle recommendations)
Other: Dietary Intervention — Receive dietary instructions
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
  Arms: Group I (diet, physical activity)
Other: Exercise Intervention — Complete aerobic and strength/resistance exercises
  Arms: Group I (diet, physical activity)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial studies the effects of a diet and physical activity intervention on blood measures of lipids and insulin resistance in patients with prostate cancer undergoing radiation therapy (RT) and androgen deprivation therapy (ADT). ADT effectively slows the growth of prostate cancer cells, thereby enhancing the therapeutic effectiveness of RT. Despite the clinical gains, ADT leads to an array of side effects including insulin resistance, abnormal lipid levels, weight gain, increased visceral fat mass coupled with increased muscle wasting, and quality of life deterioration. A diet and physical activity intervention may intercept or prevent the abrupt metabolic and physiologic changes caused by androgen deprivation therapy in prostate cancer patients receiving ADT and RT.

DETAILED DESCRIPTION:
OUTLINE:

Patients are randomized to 1 of 2 groups.

GROUP I (DIET AND PHYSICAL ACTIVITY): Patients attend 10 in-person or virtual sessions with a registered dietitian over 6 months to receive instructions on a modified DASH diet. Patients also attend 2 one-on-one sessions with an exercise psychologist to receive instruction to complete aerobic physical activity and strength/resistance training. Patients may also complete up to 21 additional supervised exercise sessions.

GROUP II (CONTROL): Patients attend a single in-person or virtual session with a registered dietitian to receive standard lifestyle recommendations based on the United States (US) dietary guidelines, activity goal of 30 minutes of physical activity 5 days/week; and discussion of the health benefits of weight maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 40 years
* Histologically confirmed adenocarcinoma of the prostate, (D'Amico risk category intermediate or high risk, localized or locoregional)
* Primary treatment is RT + ADT [Zoladex, Lupron, Degarelix, and other luteinizing hormone-releasing hormone (luteinizing hormone releasing hormone [LHRH])-directed therapies] with standard RT dose and fractionation (anti-androgen monotherapy will not be allowed
* Physically able to undertake an exercise program

Exclusion Criteria:

* Advanced, metastatic disease
* Planning to join a commercial/structured diet change or fitness program
* Have significant pre-existing T2D (poor glycemic control while on medication, defined as hemoglobin A1c of >= 10 within the prior 12 months) or significant pre-existing cardiovascular disease (CVD) (myocardial infarction or stroke within prior six months)
* Physician confirmed cognitive impairment or alcohol/narcotic abuse

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marian L. Neuhouser, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Group I (Diet, Physical Activity): Patients attend 10 in-person or virtual sessions with a registered dietitian over 6 months to receive instruction on following a healthy diet pattern. Patients also attend 2 one-on-one sessions with an exercise psychologist to receive instruction on aerobic physical activity and strength/resistance training. Patients may also complete up to 21 additional supervised exercise sessions.
  Dietary Intervention: Receive dietary instructions
  Exercise Intervention: Complete aerobic and strength/resistance exercises
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
- Group II (Standard Lifestyle Recommendations): Patients receive standard lifestyle recommendations and attend a single individual session with a dietitian to review the US dietary guidelines, activity goal of 30 minutes of physical activity 5 days/week.
Period: Overall Study
Arm/Group | Group I (Diet, Physical Activity) | Group II (Standard Lifestyle Recommendations)
Started | 9 | 11
Completed | 7 | 8
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Withdrawal due to complications with standard of care treatment | 2 | 0

BASELINE CHARACTERISTICS:
Population: Participants randomized to the intervention or control arms
Groups:
- Group I (Diet, Physical Activity): Patients attend 10 in-person or virtual sessions with a registered dietician over 6 months to receive diet instructions. Patients also attend 2 one-on-one sessions with an exercise psychologist to receive instruction to complete aerobic physical activity and strength/resistance training. Patients may also complete up to 21 additional supervised exercise sessions.
  Dietary Intervention: Receive dietary instructions
  Exercise Intervention: Complete aerobic and strength/resistance exercises
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
- Group II (Standard Lifestyle Recommendations): Patients receive standard lifestyle recommendations and attend an individual session with a dietitian over 20-30 minutes including US dietary guidelines, activity goal of 30 minutes of physical activity 5 days/week; and discussion of the health benefits of weight loss along with general behavior change suggestions for weight loss.
  Best Practice: Receive standard lifestyle recommendations
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
- Total: Total of all reporting groups
Arm/Group | Group I (Diet, Physical Activity) | Group II (Standard Lifestyle Recommendations) | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 7 | 11 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.0 (5.7) | 73.6 (4.5) | 72.43 (5.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 9 | 11 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 8 | 11 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 11 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 11 | 20

OUTCOME MEASURES:

1. Primary Outcome: Effects of the Intervention on ADT-induced Changes in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR)
Description: Data is reported as a percentage change in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) score from baseline. HOMA-IR is an index to estimate the insulin resistance of a patient. HOMA-IR is defined as (glucose (mg/dl) insulin (uIU/ml)) / 405.
Time Frame: 0 months, 6 months
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Group I (Diet, Physical Activity) | Group II (Standard Lifestyle Recommendations)
Number analyzed (Participants) | 7 | 8
percentage change | 4.5 (52.1) | 42.7 (28.1)

2. Primary Outcome: Effects of the Intervention on ADT-induced Changes in Body Weight
Description: Change in body weight from baseline.
Time Frame: 0 months, 6 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Group I (Diet, Physical Activity) | Group II (Standard Lifestyle Recommendations)
Number analyzed (Participants) | 7 | 8
kg | -1.24 (2.6) | 1.01 (1.9)

3. Primary Outcome: Effects of the Intervention on ADT-induced Changes in Waist Circumference
Description: Change in waist circumference from baseline. Waist circumference was measured at 1" above umbilicus.
Time Frame: 0 months, 6 months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Group I (Diet, Physical Activity) | Group II (Standard Lifestyle Recommendations)
Number analyzed (Participants) | 7 | 8
cm | 3.4 (1.5) | 1.8 (7.3)

4. Primary Outcome: Effects of the Intervention on ADT-induced Changes in Lean Mass
Description: Change in lean mass from baseline. Lean mass was measured by Dual-Energy X-ray Absorptiometry (DEXA).
Time Frame: 0 months, 6 months
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Group I (Diet, Physical Activity) | Group II (Standard Lifestyle Recommendations)
Number analyzed (Participants) | 7 | 8
g | -998 (1604) | -1129 (1423)

5. Primary Outcome: Effects of the Intervention on ADT-induced Changes in Fat Mass
Description: Change in fat mass from baseline. Fat mass was measured by Dual-Energy X-ray Absorptiometry (DEXA).
Time Frame: 0 months, 6 months
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Group I (Diet, Physical Activity) | Group II (Standard Lifestyle Recommendations)
Number analyzed (Participants) | 7 | 8
g | 1307 (2984) | 2491 (1189)

ADVERSE EVENTS:
Time Frame: up to 6 months
Arm/Group | Group I (Diet, Physical Activity) | Group II (Standard Lifestyle Recommendations)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 5/9 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (Diet, Physical Activity) (N=9) | Group II (Standard Lifestyle Recommendations) (N=11)
Knee Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Hip and back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
elevated liver function tests (Hepatobiliary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Presyncope (Cardiac disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This is a pilot feasibility study with a sample size of 20 participants. Results should be interpreted accordingly.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-03): https://cdn.clinicaltrials.gov/large-docs/15/NCT04870515/Prot_SAP_001.pdf
  • Informed Consent Form (2022-05-07): https://cdn.clinicaltrials.gov/large-docs/15/NCT04870515/ICF_000.pdf